CLINICAL TRIAL: NCT01569152
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Worldwide, Dose-Ranging Clinical Trial With a Proof-of-Concept Lead Cohort to Evaluate the Safety, Tolerability, and Efficacy of MK-8457 + MTX in Patients With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: Safety and Efficacy of MK-8457 and Methotrexate (MTX) in Participants With Active Rheumatoid Arthritis Despite MTX Therapy (P08683, MK-8457-008)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P08683; MK-8457-008 (Other: Merck); 2012-000439-17 (EudraCT Number); 132235 (Registry Identifier: JAPIC-CTI); P08683 (Other: Merck)
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Base Study Phase IIa: MK-8457 (Experimental): Participants received MK-8457 100 mg dosed twice daily (BID) orally with MTX at the stable dose received upon study enrollment. Phase IIa lasted up to 24 weeks.
  Interventions: Drug: MK-8457 100 mg; Drug: Methotrexate
- Base Study Phase IIa: Placebo (Placebo Comparator): Participants received placebo dosed BID orally with MTX at the stable dose received upon study enrollment. Phase IIa lasted up to 24 weeks.
  Interventions: Drug: Dose-Matched Placebo; Drug: Methotrexate
- Safety Extension Period 3: MK-8457 (Experimental): Participants received MK-8457 100 mg BID orally with MTX at the stable dose received upon study enrollment. Period 3 was to last up to 2 years.
  Interventions: Drug: MK-8457 100 mg; Drug: Methotrexate

INTERVENTIONS:
Drug: MK-8457 100 mg — MK-8457 100 mg dosed orally BID
  Arms: Base Study Phase IIa: MK-8457; Safety Extension Period 3: MK-8457
Drug: Dose-Matched Placebo — Dose-matched placebo dosed orally BID
  Arms: Base Study Phase IIa: Placebo
Drug: Methotrexate — MTX dosed at the stable dose receive upon study entry
  Other Names: MTX

SUMMARY:
The purpose of this study is to assess the safety and efficacy of MK-8457 + Methotrexate (MTX) in participants with active rheumatoid arthritis (RA) despite MTX therapy. The primary hypothesis is that at least 1 dose of MK-8457 + MTX will be superior to placebo + MTX as measured by the percentage of participants who achieve American College of Rheumatology 20 (ACR 20) response after 12 weeks of treatment.

DETAILED DESCRIPTION:
In Base Study Phase IIa, participants were to receive blinded MK-8457 100 mg or matched placebo for up to 24 weeks. At Week 12 and 18 of Phase IIa, efficacy evaluation was conducted to assess eligibility for early escape, defined as <20% reduction in both tender and swollen joint counts. The study plan included Base Study Phase IIb in which dose range finding or dose-response was to be evaluated, depending on the outcome of Phase IIa. Participants who completed Phase IIa or Phase IIb and those eligible for early escape could enroll in Period 3, a 2-year Safety Extension.

All participants must have been treated with MTX for at least 3 months prior to screening and have been receiving a stable dose of MTX for at least 4 weeks prior to screening.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis for at least 6 months prior to screening
* Active rheumatoid arthritis as defined by the presence of >= 6 swollen joints (of 66 count) and >= 6 tender joints (of 68 joint count)
* C-reactive protein blood level >0.9 mg/dL
* Anti-citrullinated protein antibody positive and/or rheumatoid factor positive at screening
* American College of Rheumatology Functional Class I, II, or III
* Received methotrexate for a minimum of 3 months prior to screening with a regionally appropriate stable weekly dose for at least 4 weeks prior to screening
* If using oral corticosteroids, the participant must be on a stable dose of 10 mg prednisone
* No history of either untreated, latent, or active tuberculosis prior to baseline
* Participants of reproductive potential must agree to remain abstinent or use 2 acceptable methods of birth control

Exclusion Criteria:

* Presence of inflammatory disease other than rheumatoid arthritis, including but not limited to psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus, or Lyme disease
* Positive hepatitis B surface antigen or hepatitis C test result or the presence of Human immunodeficiency virus (HIV) infection
* HIV positive
* User of recreational or illicit drugs or has had a history (within the previous 2 years) of drug or alcohol abuse or dependence
* Females of childbearing potential who are pregnant, intend to become pregnant, or are lactating;
* Severe opportunistic infection within 6 months prior to study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-05-22 (Actual); Primary Completion 2013-10-03 (Actual); Study Completion 2013-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 58 trial centers in the United States, Canada, Chile, Denmark, South Africa, Germany, Hungary, Japan, Lithuania, Moldova, Poland, South Korea, Taiwan, and in the United Kingdom. A total of 213 participants were screened and 82 were enrolled.
Pre-assignment Details: The internal data monitoring committee made the decision to discontinue the study before initiation of Base Study Phase IIb. Thus, participants were enrolled in Base Study Phase IIa and the Study Extension (Period 3) only.
Groups:
- Base Study Phase IIa: MK-8457: MK-8457 100mg BID + MTX for up to 24 weeks in Base Study Phase IIa
- Base Study Phase IIa: Placebo: Placebo + MTX for up to 24 weeks in Base Study Phase IIa
- Safety Extension Period 3: MK-8457: MK-8457 100 mg BID + MTX for up to approximately 52 weeks in Safety Extension Period 3. Participants who completed or had early escape from Base Study Phase IIa were eligible to enroll in Safety Extension Period 3.
Period: Phase IIa, Period 1
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo | Safety Extension Period 3: MK-8457
Started | 41 | 41 | 0
Completed | 20 | 9 | 0
Not Completed | 21 | 32 | 0
Not completed — Early Escape | 5 | 22 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 9 | 8 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Period: Safety Extension, Period 3
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo | Safety Extension Period 3: MK-8457
Started | 0 | 0 | 55 (Includes 29 completers and 26 early escapees from Base Study Phase IIa)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 55
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Study terminated by Sponsor | 0 | 0 | 47

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 31 | 66
  >=65 years | 6 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (9.5) | 56.1 (11.1) | 54.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 63
  Male | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an American College of Rheumatology (ACR) 20 Response at Week 12
Description: ACR responses are numerical measurements of improvement in multiple disease assessment criteria. An ACR20 response is defined as a ≥20% improvement in 1) swollen joint count (66 joints) and tender joint count (68 joints) (0 = Absent; 1 = Present) and 2) ≥20% improvement in 3 of the following 5 assessments: a) a participant's overall assessment of pain on a visual analog scale (VAS, no pain =0 to extreme pain =100); b) Patient's Global Assessment of Disease Activity VAS (doing very well =0 to doing very poor =100); c) Investigator's Global Assessment of Disease Activity VAS (doing very well =0 to doing very poor =100 ; d) participant's assessment of function across 8 functional areas as measured by Health Assessment Questionnaire (HAQ), total scores ranging from no difficulty =0 to inability to perform tasks =24; and e) serum C-Reactive Protein (decrease indicates improvement). This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline ACR20 measurement (last observation carried forward)
Measure: Number; unit: Percentage of participants
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 41 | 41
Percentage of participants | 68.29 | 24.39
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference of percentages = 43.90, 95% CI 2-sided [24.52 to 63.28]

2. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28) as Measured by Erythrocyte Sedimentation Rate (ESR) at Week 12
Description: The DAS28-ESR is a continuous parameter based upon a statistically-derived index combining tender joints (28 joints, TEN28), swollen joints (28 joints, SW28), ESR (an inflammatory marker), and Patient's Global Assessment of Disease Activity VAS (GH). It is defined as follows: DAS28-ESR = 0.56 × SQRT(TEN28) + 0.28 × SQRT(SW28) + 0.70 × ln (ESR) + 0.014 × GH. SQRT = square root. The DAS28-ESR is a scale ranging from 0 to 10 with higher values indicating greater rheumatoid arthritis (RA) disease activity. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had both Baseline and Week 12 DAS28-ESR measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 37 | 39
Units on a scale | -2.00 [-2.40 to -1.61] | -1.02 [-1.41 to -0.64]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in least squares means = -0.98, 95% CI 2-sided [-1.53 to -0.43]

3. Secondary Outcome: Change From Baseline in DAS28 as Measured by C-Reactive Protein (CRP) at Week 12
Description: The DAS28-CRP is a continuous parameter based upon a statistically-derived index combining tender joints (28 joints, TEN28), swollen joints (28 joints, SW28), CRP (an inflammatory marker), and Patient's Global Assessment of Disease Activity VAS (GH). It is defined as follows: DAS28-CRP = 0.56 × SQRT(TEN28) + 0.28 × SQRT(SW28) + 0.36 × ln (CRP+1) + 0.014 × GH + 0.96. The DAS28-CRP is a scale ranging from 0 to 10 with higher values indicating greater RA disease activity. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had both Baseline and Week 12 DAS28-CRP measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 37 | 39
Units on a scale | -1.98 [-2.34 to -1.61] | -0.87 [-1.23 to -0.51]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in least squares means = -1.11, 95% CI 2-sided [-1.62 to -0.60]

4. Secondary Outcome: Percentage of Participants Achieving an ACR70 Response at Week 12
Description: ACR responses are numerical measurements of improvement in multiple disease assessment criteria. An ACR70 response is defined as a ≥70% improvement in 1) swollen joint count (66 joints) and tender joint count (68 joints) (0 = Absent; 1 = Present) and 2) ≥70% improvement in 3 of the following 5 assessments: a) a participant's overall assessment of pain on a visual analog scale (VAS, no pain =0 to extreme pain =100); b) Patient's Global Assessment of Disease Activity VAS (doing very well =0 to doing very poor =100); c) Investigator's Global Assessment of Disease Activity VAS (doing very well =0 to doing very poor =100 ; d) participant's assessment of function across 8 functional areas as measured by Health Assessment Questionnaire (HAQ), total scores ranging from no difficulty =0 to inability to perform tasks =24; and e) serum C-Reactive Protein (decrease indicates improvement). This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline ACR70 measurement
Measure: Number; unit: Percentage of participants
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 41 | 41
Percentage of participants | 19.51 | 4.88
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p = 0.044, Cochran-Mantel-Haenszel; Difference in percentages = 14.63, 95% CI 2-sided [0.83 to 28.44]

5. Secondary Outcome: Percentage of Participants Achieving Hybrid ACR Response at Week 12
Description: Hybrid ACR Response evaluates the improvement in active RA by combining elements of the ACR20/50/70 with a categorical score of the mean change in the core set measures (tender joint count, swollen joint count, Patient's Global Assessment of Disease Activity, Investigator's Global Assessment of Disease Activity, disability index of the HAQ, and CRP). The mean percentage improvement from Baseline in the core set measures was computed and used with the participant's ACR20, ACR50, and ACR70 status to determine the hybrid ACR response in a lookup table. The range of values was -100 to 100, with a positive change indicating improvement. This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: Due to the early termination of the study, analysis for this outcome measure was not performed according to the protocol because complete data were not available.
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants Achieving an ACR-N Response at Week 12
Description: The ACR-N response is the minimum of the following: 1) the percent decrease from Baseline in tender joint counts (68 joints, 0 = absent, 1 = present); 2) the percent decrease from Baseline in swollen joint counts (66 joints, 0 = absent, 1 = present); and 3) the median percent decrease from Baseline for the following: a) Patient's Global Assessment of Pain (VAS, 0 mm = "no pain" and 100 mm = "extreme pain"); b) Patient's Global Assessment of Disease Activity (VAS, 0 mm = doing very well to 100 mm = doing very poor); c) Investigator's Global Assessment of Disease Activity (VAS, 0 mm = doing very well to 100 mm = doing very poor); d. physical function as measured by the HAQ (Likert scale, 0 to 3 with a lower score indicating less disability); and e) CRP. This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: as for outcome 5
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants Achieving a DAS28-ESR Response at Week 12
Description: The DAS28-ESR is a continuous parameter based upon a statistically-derived index combining tender joints (28 joints, TEN28), swollen joints (28 joints, SW28), ESR, and Patient's Global Assessment of Disease Activity VAS (GH). It is defined as follows: DAS28-ESR = 0.56 × SQRT(TEN28) + 0.28 × SQRT(SW28) + 0.70 × ln (ESR) + 0.014 × GH. SQRT = square root. The DAS28-ESR is a scale ranging from 0 to 10 with higher values indicating greater RA disease activity. Depending upon the DAS28-ESR value for a given visit, change in DAS28-ESR is categorized as follows: No Response (reduction from Baseline ≤0.6), No response or Moderate Response (reduction >0.6 - 1.2), and Moderate or Good Response (reduction >1.2). The percentage of participants with a Moderate or Good change in DAS28-ESR was reported. This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline DAS28-ESR measurement
Measure: Number; unit: Percentage of participants
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 41 | 41
Percentage of participants | 70.73 | 39.02
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; Difference in percentages = 31.71, 95% CI 2-sided [11.29 to 52.13]

8. Secondary Outcome: Percentage of Participants Achieving a DAS28-CRP Response at Week 12
Description: The DAS28-CRP is a continuous parameter based upon a statistically-derived index combining tender joints (28 joints, TEN28), swollen joints (28 joints, SW28), CRP, and Patient's Global Assessment of Disease Activity VAS (GH). It is defined as follows: DAS28-CRP = 0.56 × SQRT(TEN28) + 0.28 × SQRT(SW28) + 0.36 × ln (CRP+1) + 0.014 × GH + 0.96. The DAS28-CRP is a scale ranging from 0 to 10 with higher values indicating greater RA disease activity. Depending upon the DAS28-CRP value for a given visit, change in DAS28-CRP is categorized as follows: No Response (reduction from Baseline ≤0.6), No response or Moderate Response (reduction >0.6 - 1.2), and Moderate or Good Response (reduction >1.2). The percentage of participants with a Moderate or Good change in DAS28-CRP was reported. This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline DAS28-CRP measurement
Measure: Number; unit: Percentage of participants
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 41 | 41
Percentage of participants | 73.17 | 43.90
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel; Difference in percentages = 29.27, 95% CI 2-sided [8.90 to 49.63]

9. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR Remission at Week 12
Description: The DAS28-ESR is a continuous parameter based upon a statistically-derived index combining tender joints (28 joints, TEN28), swollen joints (28 joints, SW28), ESR, and Patient's Global Assessment of Disease Activity VAS (GH). It is defined as follows: DAS28-ESR = 0.56 × SQRT(TEN28) + 0.28 × SQRT(SW28) + 0.70 × ln (ESR) + 0.014 × GH. SQRT = square root. The DAS28-ESR is a scale ranging from 0 to 10 with higher values indicating greater RA disease activity. DAS28-ESR remission is defined as a value <2.6 at the visit. This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 41 | 41
Percentage of participants | 9.76 | 0
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p = 0.039, Cochran-Mantel-Haenszel; Difference in percentages = 9.76, 95% CI 2-sided [0.67 to 18.84]

10. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP Remission at Week 12
Description: The DAS28-CRP is a continuous parameter derived from the formula: 0.56 × the square root of the tender joint count (0-28) + 0.28 × the square root of the swelling joint count (0-28) + 0.36 × the C reactive protein value (in mg/L +1) + 0.014 × Patient's Global Assessment of Disease Activity VAS of 0-100 mm + 0.96. The DAS28-CRP is a scale ranging from 0 to 10 with higher values indicating greater RA disease activity. DAS28-CRP remission is defined as a value <2.6 at the visit. This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 41 | 41
Percentage of participants | 12.20 | 0.00
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel; Difference in percentages = 12.20, 95% CI 2-sided [2.18 to 22.21]

11. Secondary Outcome: DAS28-ESR Area Under the Curve (AUC)
Description: DAS28-ESR AUC was to be calculated from the DAS28-ESR score versus time curve, which provided an assessment of changes in disease activity over time. The DAS28-ESR AUC was to be calculated using the trapezoidal rule as the DAS28-ESR multiplied by the duration of the assessment period (in weeks) and was to be expressed as %-weeks. A higher calculated AUC value indicates higher disease activity (worse). This outcome measure applied to Base Study participants only.
Time Frame: Up to 12 weeks
Population: as for outcome 5
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: DAS28-CRP Area Under the Curve (AUC)
Description: DAS28-CRP AUC was to be calculated from the DAS28-CRP score versus time curve, which provided an assessment of changes in disease activity over time. The DAS28-CRP AUC was to be calculated using the trapezoidal rule as the DAS28-CRP multiplied by the duration of the assessment period (in weeks) and was to be expressed as %-weeks. A higher calculated AUC value indicates higher disease activity (worse). This outcome measure applied to Base Study participants only.
Time Frame: Up to 12 weeks
Population: as for outcome 5
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Tender Joint Count at Week 12
Description: Tender Joint Count was examined on 68 joints of the fingers, elbows, hips, knees, ankles, and toes distal for pain in response to pressure or passive motion at the study time points. Joint pain was scored as 0 = Absent; 1 = Present for each joint. The overall Tender Joint Count ranged from 0 to 68. A higher score indicated greater disease severity. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline tender joint count
Measure: Least Squares Mean (95% Confidence Interval); unit: Tender joints
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 38 | 39
Tender joints | -13.53 [-16.73 to -10.34] | -8.78 [-11.96 to -5.60]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p = 0.028, Constrained Longitudinal Data Analysis; Difference in least squares means = -4.75, 95% CI 2-sided [-8.99 to -0.52]

14. Secondary Outcome: Change From Baseline in Swollen Joint Count at Week 12
Description: Swollen joint count included 66 joints (same joints as for tender joint count except this excluded evaluation of hips) that were assessed for the presence of swelling. Soft tissue swelling was considered to be present if there was palpable or visible evidence of capsular distention considered to be due to either synovial thickening and/or a joint effusion. Bony swelling, nodule formation, and joint deformity were excluded from consideration. A swollen joint was scored as 0 = Absent; 1 = Present for each joint. The overall swollen joint count ranged from 0 to 66. A higher score indicated greater disease severity. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline swollen joint count
Measure: Least Squares Mean (95% Confidence Interval); unit: Swollen joints
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 38 | 39
Swollen joints | -10.29 [-13.01 to -7.58] | -7.65 [-10.34 to -4.95]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p = 0.110, Constrained Longitudinal Data Analysis; Difference in least squares means = -2.65, 95% CI 2-sided [-5.91 to 0.62]

15. Secondary Outcome: Change From Baseline in the Simplified Disease Activity Index (SDAI) at Week 12
Description: SDAI is the simple linear sum of the following parameters: tender joint count (TJC) and swollen joint count (SJC) based on a 28-joint assessment, Patient's Global Assessment of Disease Activity [PGA, VAS 0 to 10 cm], Investigator's Global Assessment of Disease Activity (MDGA, VAS 0 to 10 cm) and CRP levels (mg/dL). SDAI =TJC + SJC + PGA + MDGA + CRP. Overall scores can range from 0.0 to 86.0. A higher score indicated greater disease severity. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline SDAI assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 37 | 39
Units on a scale | -23.73 [-28.50 to -18.96] | -13.17 [-17.90 to -8.45]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p = 0.002, Constrained Longitudinal Data Analysis; Difference in least squares means = -10.56, 95% CI 2-sided [-16.97 to -4.15]

16. Secondary Outcome: Change From Baseline in the Short Form Health Survey (SF-36) at Week 12
Description: The SF-36 is a health-related quality of life instrument that consists of 8 multi-item scales: limitations in physical functioning due to health problems, limitations in usual role activities due to physical health problems, bodily pain, general mental health (psychological distress and well-being), limitations in usual role activities due to personal or emotional problems, limitations in social functioning due to physical or mental health problems, vitality (energy and fatigue), and general health perception. Each scale is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. The lower the score the greater the disability i.e., a score of 0 corresponds to maximum disability and a score of 100 corresponds to no disability. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) at Week 12
Description: The FACIT-F is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). The higher the participant's response to the questions the greater the participant's fatigue. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change From Baseline in the Patient's Global Assessment of Disease Status/Activity (PGADSA) at Week 12
Description: A participant's overall assessment of pain was assessed from the amount of pain due to arthritis experienced during the past 48 hours on a VAS, where 0 mm = doing very well to 100 mm = doing very poor. A negative change from Baseline indicates improvement. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline PGADSA assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 37 | 39
Units on a scale | -29.06 [-35.93 to -22.19] | -8.21 [-15.00 to -1.43]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in least squares means = -20.84, 95% CI 2-sided [-29.98 to -11.71]

19. Secondary Outcome: Change From Baseline in the Investigator's Global Assessment of Disease Status/Activity (IGADSA) at Week 12
Description: The Investigator's Global Assessment of Disease Status/Activity (IGADSA) is measured with scores ranging from 0 to 100 mm (VAS, 0 mm = doing very well to 100 mm = doing very poor). A negative change from Baseline indicates improvement. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline IGADSA assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 38 | 39
Units on a scale | -34.21 [-41.80 to -26.63] | -14.73 [-22.23 to -7.23]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in least squares means = -19.48, 95% CI 2-sided [-29.69 to -9.28]

20. Secondary Outcome: Change From Baseline in the Patient's Global Assessment of Pain (PGAP) at Week 12
Description: A participant's overall assessment of pain was assessed from the amount of pain due to arthritis experienced during the past 48 hours on a VAS where 0 mm = "no pain" and 100 mm = "extreme pain". A negative change from Baseline indicates improvement. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline PGAP assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 37 | 39
Units on a scale | -28.85 [-37.17 to -20.54] | -8.17 [-16.42 to 0.09]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in least squares means = -20.69, 95% CI 2-sided [-31.29 to -10.09]

21. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire Disability (HAQ Disability Index) at Week 12
Description: The functional status of the participant was assessed using the Disability Index of the HAQ on a Likert scale. This 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area. The overall score for the Disability Index is the mean of the 8 functional area scores and also ranges from 0 to 3, with a lower score indicating less disability. A negative change from Baseline indicates improvement. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline HAQ Disability Index assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 38 | 39
Units on a scale | -0.67 [-0.83 to -0.51] | -0.05 [-0.21 to 0.11]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in least squares means = -0.62, 95% CI 2-sided [-0.84 to -0.40]

22. Secondary Outcome: Change From Baseline in Serum C-Reactive Protein (CRP) at Week 12
Description: C-Reactive Protein is an inflammatory marker with a normal reference range of less than 0.9 mg/dL. Change from Baseline in CRP at Week 12 (Week 12 concentration minus Baseline concentration). This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline serum CRP assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 38 | 39
mg/dL | -0.76 (0.83) [-1.66 to 0.14] | 0.83 (0.86) [-0.07 to 1.73]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p = 0.007, Constrained Longitudinal Data Analysis; Difference in least squares means = -1.59, 95% CI 2-sided [-2.73 to -0.45]

23. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 12
Description: The ESR is the rate at which red blood cells sediment in a period of one hour, and is a non-specific measure of inflammation. Change from Baseline is ESR at Week 12 minus ESR at Baseline. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline ESR assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: mm/hr
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 38 | 39
mm/hr | -6.80 [-13.98 to 0.38] | -1.90 [-9.03 to 5.23]
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p = 0.315, Constrained Longitudinal Data Analysis; Difference in least squares means = -4.90, 95% CI 2-sided [-14.54 to 4.74]

24. Secondary Outcome: Change From Baseline in Hemoglobin at Week 12
Description: Hemoglobin is the iron-containing oxygen-transport metalloprotein in red blood cells. Change from Baseline is hemoglobin at Week 12 minus hemoglobin at Baseline. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had non-missing Baseline and Week 12 hemoglobin values
Measure: Mean (Standard Deviation); unit: gm/dL
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 39 | 39
gm/dL | 0.11 (0.83) | -0.07 (0.86)

25. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response at Week 12
Description: ACR responses are numerical measurements of improvement in multiple disease assessment criteria. An ACR50 response is defined as a ≥50% improvement in 1) swollen joint count (66 joints) and tender joint count (68 joints) (0 = Absent; 1 = Present) and 2) ≥50% improvement in 3 of the following 5 assessments: a) a participant's overall assessment of pain on a visual analog scale (VAS, no pain =0 to extreme pain =100); b) Patient's Global Assessment of Disease Activity VAS (doing very well =0 to doing very poor =100); c) Investigator's Global Assessment of Disease Activity VAS (doing very well =0 to doing very poor =100 ; d) participant's assessment of function across 8 functional areas as measured by Health Assessment Questionnaire (HAQ), total scores ranging from no difficulty =0 to inability to perform tasks =24; and e) serum C-Reactive Protein (decrease indicates improvement). This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline ACR50 assessment
Measure: Number; unit: Percentage of participants
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 41 | 41
Percentage of participants | 36.59 | 4.88
Statistical Analysis 1: Comparison: Base Study Phase IIa: MK-8457 vs Base Study Phase IIa: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentages = 31.71, 95% CI 2-sided [15.56 to 47.86]

26. Secondary Outcome: Percentage of Participants With an ACR20 Response Over Time
Description: as for outcome 1
Time Frame: Week 1, Week 2, Week 4, Week 6, Week 18 and Week 24
Population: Randomized participants in Base Study Phase IIa who received at least one dose of study drug and had at least one post-baseline ACR20 measurement
Measure: Number; unit: Percentage of participants
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo
Number analyzed (Participants) | 41 | 41
Percentage of participants
  Week 1 | 12.2 | 9.8
  Week 2 | 51.2 | 14.6
  Week 4 | 61.0 | 22.0
  Week 6 | 63.4 | 14.6
  Week 12 | 68.3 | 24.4
  Week 18 | 53.7 | 12.2
  Week 24 | 48.8 | 22.0

ADVERSE EVENTS:
Time Frame: Base Study Phase IIa: up to 24 weeks; Safety Extension Period 3: up to approximately 52 weeks
Arm/Group | Base Study Phase IIa: MK-8457 | Base Study Phase IIa: Placebo | Safety Extension Period 3: MK-8457
Serious Adverse Events (participants affected / at risk) | 2/41 | 0/41 | 3/55
Other Adverse Events (participants affected / at risk) | 15/41 | 9/41 | 11/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study Phase IIa: MK-8457 (N=41) | Base Study Phase IIa: Placebo (N=41) | Safety Extension Period 3: MK-8457 (N=55)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study Phase IIa: MK-8457 (N=41) | Base Study Phase IIa: Placebo (N=41) | Safety Extension Period 3: MK-8457 (N=55)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early (12 September 2013) based on preliminary analysis of data. The results of this study need to be interpreted with caution given the small sample size (82 participants) resulting from the early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.